CLINICAL TRIAL: NCT03511001
Title: Effects Among Smokers Who Use and Do Not Use E-Cigarettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California State University, San Marcos (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1119341-85085; 1SC3GM122628 (NIH)
Record Dates: First submitted 2018-04-10; First posted 2018-04-27 (Actual); Results first posted 2021-09-05 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-08

CONDITIONS: Toxicant Exposure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-Cigarette (Experimental): 6 weeks of JUUL electronic cigarettes
  Interventions: Other: E-Cigarette Vs. Smoking as Usual
- Assessment Only (Active Comparator): 6 weeks of smoking as usual
  Interventions: Other: E-Cigarette Vs. Smoking as Usual

INTERVENTIONS:
Other: E-Cigarette Vs. Smoking as Usual — 6 weeks of JUUL e-cigarettes vs. 6 weeks of smoking as usual

SUMMARY:
This study compares effects among Latino and African American cigarette smokers who use e-cigarettes with those who continue smoking as usual.

ELIGIBILITY:
Inclusion Criteria:

* > 21 years of age
* Smoked cigarettes on > 25 of past 30 days
* Smoked > 5 cigarettes per day on days smoked
* Smoked cigarettes > 6 months
* Carbon monoxide > 5 PPM at baseline
* Hispanic/Latino or African American/Black
* Fluent in English or Spanish
* Willing to switch from smoking cigarettes to ECs for 6 weeks
* Regular access to telephone
* Transportation to attend appointments (KC Only)

Exclusion Criteria:

* Primary use of other tobacco products or equal use of cigarettes and other tobacco products
* Electronic cigarette use on > 4 of the past 30 days
* Currently in a smoking cessation program or another clinical trial
* Use of nicotine replacement therapy or medication which aids smoking cessation in the past 30 days
* Hospitalization for a psychiatric issue in the past 30 days
* Heart-related event in the past 30 days. Examples include heart attack, stroke, severe angina (i.e. chest pain), ischemic heart disease, and vascular disease
* Uncontrolled blood pressure at baseline
* Planning to move out of San Diego or Kansas City in the next 6 weeks
* Another person in the household enrolled in the study
* Women: pregnant, breastfeeding, or planning to become pregnant in the next six months
* Unstable mental status or health status

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Pulvers, PhD, MPH, Principal Investigator — Associate Professor
Locations (2):
- United States (2):
  - California State University San Marcos, San Marcos, California
  - Swope Health Central, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nollen NL, Leavens ELS, Ahluwalia JS, Rice M, Mayo MS, Pulvers K. Menthol versus non-menthol flavouring and switching to e-cigarettes in black and Latinx adult menthol combustible cigarette smokers: secondary analyses from a randomised clinical trial. Tob Control. 2023 Nov;32(6):786-789. doi: 10.1136/tobaccocontrol-2021-057180. Epub 2022 Mar 29. PMID 35351805
- [Derived] Pulvers K, Rice M, Ahluwalia JS, Arnold MJ, Marez C, Nollen NL. "It is the One Thing that has Worked": facilitators and barriers to switching to nicotine salt pod system e-cigarettes among African American and Latinx people who smoke: a content analysis. Harm Reduct J. 2021 Sep 16;18(1):98. doi: 10.1186/s12954-021-00543-y. PMID 34530834
- [Derived] Arnold MJ, Nollen NL, Mayo MS, Ahluwalia JS, Leavens EL, Zhang G, Rice M, Pulvers K. Harm Reduction Associated with Dual Use of Cigarettes and e-Cigarettes in Black and Latino Smokers: Secondary Analyses from a Randomized Controlled e-Cigarette Switching Trial. Nicotine Tob Res. 2021 Oct 7;23(11):1972-1976. doi: 10.1093/ntr/ntab069. PMID 33837422
- [Derived] Pulvers K, Nollen NL, Rice M, Schmid CH, Qu K, Benowitz NL, Ahluwalia JS. Effect of Pod e-Cigarettes vs Cigarettes on Carcinogen Exposure Among African American and Latinx Smokers: A Randomized Clinical Trial. JAMA Netw Open. 2020 Nov 2;3(11):e2026324. doi: 10.1001/jamanetworkopen.2020.26324. PMID 33206193

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | E-Cigarette | Assessment Only
Started | 126 | 61
Completers Analyzed | 114 (1 participant was excluded post-randomization due to not meeting race/ethnicity inclusion criteria.) | 61
Completed | 115 | 54
Not Completed | 11 | 7

BASELINE CHARACTERISTICS:
Population: One post-randomization exclusion from analyses due to not meeting race/ethnicity inclusion criteria
Groups:
- Total: Total of all reporting groups
Arm/Group | E-Cigarette | Assessment Only | Total
Number analyzed (Participants) | 125 | 61 | 186
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.1 (12.7) | 41.7 (11.9) | 43.3 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 26 | 75
  Male | 76 | 35 | 111
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 63 | 31 | 94
  Not Hispanic or Latino | 62 | 30 | 92
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 4 | 12
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 66 | 30 | 96
  White | 36 | 24 | 60
  More than one race | 9 | 2 | 11
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 125 | 61 | 186
High school education or less [Count of Participants; unit: Participants] | 68 | 34 | 102
200% federal poverty level or lower [Count of Participants; unit: Participants] | 93 | 45 | 138
Never married [Count of Participants; unit: Participants] | 59 | 31 | 90
Menthol smoker [Count of Participants; unit: Participants] | 68 | 34 | 102
Duration smoking in years [Mean (Standard Deviation); unit: years] | 17.5 (12.8) | 15.5 (12.5) | 16.8 (12.7)
Time to first cigarette 30 minutes or less [Count of Participants; unit: Participants] — Participants were asked how soon after waking they typically smoked first cigarette of the day. Response options included within 30 minutes of waking or after 30 minutes of waking.
  Participants | 91 | 44 | 135
Days smoked in past 7 days [Mean (Standard Deviation); unit: days] | 6.9 (0.5) | 6.7 (0.9) | 6.8 (0.6)
Cigarettes per day in past 7 days [Mean (Standard Deviation); unit: cigarettes per day] | 12.4 (7.7) | 11.5 (6.1) | 12.1 (7.2)
Days used e-cigarettes in past 7 days [Mean (Standard Deviation); unit: days] | 0.03 (0.28) | 0.08 (0.33) | 0.05 (0.30)
E-cigarette uses in past 7 days [Mean (Standard Deviation); unit: uses per day] | 0.05 (0.48) | 0.09 (0.36) | 0.06 (0.45)
History of chronic obstructive pulmonary disorder [Count of Participants; unit: Participants] | 10 | 0 | 10
History of asthma [Count of Participants; unit: Participants] | 31 | 10 | 41
History of mental health diagnosis [Count of Participants; unit: Participants] | 77 | 30 | 107
History of substance abuse [Count of Participants; unit: Participants] | 64 | 24 | 88
Urine cotinine, ng/mL [Median (Inter-Quartile Range); unit: ng/mL] | 928 [463 to 1476] | 1061 [534 to 1720] | 998 [480 to 1653]
Urine NNAL, pg/mL [Median (Inter-Quartile Range); unit: pg/mL] | 124 [45 to 197] | 88 [58 to 197] | 110 [52 to 197]
Carbon monoxide, ppm [Median (Inter-Quartile Range); unit: ppm] | 16 [11 to 22] | 17 [11 to 25] | 17 [11 to 23]
Lung function, FEF 25%-75%, L/s [Median (Inter-Quartile Range); unit: L/s] | 3.0 [2.1 to 4.1] | 2.8 [2.1 to 4.0] | 3.0 [2.1 to 4.1]
Respiratory symptoms, number [Median (Inter-Quartile Range); unit: units on a scale] — American Thoracic Society Questionnaire total score ranges from 0-32; higher scores reflect worse outcomes
  units on a scale | 11 [5 to 18] | 8 [4 to 13] | 10 [5 to 17]
Systolic blood pressure [Median (Inter-Quartile Range); unit: mm Hg] | 130 [115 to 142] | 129 [118 to 140] | 129 [116 to 142]
Diastolic blood pressure [Median (Inter-Quartile Range); unit: mm Hg] | 81 [76 to 89] | 83 [74 to 88] | 82 [76 to 89]

OUTCOME MEASURES:

1. Primary Outcome: Toxicant Exposure
Description: Urinary NNAL at week 6. Urinary NNAL measured by liquid chromatography-tandem mass spectrometry (LC-MS/MS)
Time Frame: 6 weeks
Population: Of the 115 participants enrolled in the treatment group, one was excluded post-randomization due to not meeting race/ethnicity inclusion criteria. Total number analyzed in treatment group was 114.
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | E-Cigarette | Assessment Only
Number analyzed (Participants) | 114 | 54
pg/ml | 40 [12 to 101] | 97 [39 to 222]

2. Secondary Outcome: Carbon Monoxide
Description: Carbon monoxide at week 6. Breath test (PPM)
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ppm
Arm/Group | E-Cigarette | Assessment Only
Number analyzed (Participants) | 114 | 54
ppm | 7 [3 to 14] | 16 [9 to 25]

3. Secondary Outcome: Respiratory Symptoms
Description: Respiratory symptoms at week 6. American Thoracic Society Questionnaire total score ranges from 0-32; higher scores reflect worse outcomes
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | E-Cigarette | Assessment Only
Number analyzed (Participants) | 114 | 54
score on a scale | 7 [3 to 12] | 9 [4 to 16]

4. Secondary Outcome: Lung Function
Description: FEF 25%-75%, L/s at week 6 measured by spirometer
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: L/sec
Arm/Group | E-Cigarette | Assessment Only
Number analyzed (Participants) | 114 | 54
L/sec | 2.8 [1.8 to 4.1] | 2.7 [2.1 to 4.1]

5. Secondary Outcome: Systolic Blood Pressure
Description: Systolic blood pressure at week 6
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | E-Cigarette | Assessment Only
Number analyzed (Participants) | 114 | 54
mmHg | 128 [117 to 142] | 133 [122 to 143]

6. Secondary Outcome: Diastolic Blood Pressure
Description: Diastolic blood pressure at week 6
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | E-Cigarette | Assessment Only
Number analyzed (Participants) | 114 | 54
mmHg | 83 [74 to 89] | 83 [75 to 89]

7. Secondary Outcome: Tobacco Dependence
Description: Tobacco dependence at week 6. Validated questions from PATH; total score ranges from 15-76, higher scores reflect worse outcomes
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | E-Cigarette | Assessment Only
Number analyzed (Participants) | 114 | 54
score on a scale | 18.5 [15.0 to 36.3] | 41.0 [33.8 to 57.5]

8. Secondary Outcome: Self-efficacy to Resist Smoking
Description: Self-efficacy to resist smoking at week 6. Brief Self Efficacy to Resist Smoking Cigarettes Scale; total score ranges from 0-60, higher score reflects better outcome
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | E-Cigarette | Assessment Only
Number analyzed (Participants) | 114 | 54
score on a scale | 43.0 [26.5 to 56.0] | 20.0 [12.5 to 30.5]

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | E-Cigarette | Assessment Only
All-Cause Mortality (participants affected / at risk) | 0/114 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/114 | 0/54
Other Adverse Events (participants affected / at risk) | 46/114 | 22/54
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | E-Cigarette (N=114) | Assessment Only (N=54)
Dry Mouth/Throat (Respiratory, thoracic and mediastinal disorders) | 46 (46) | 22 (22)
Irritated Mouth/Throat (Respiratory, thoracic and mediastinal disorders) | 24 (24) | 11 (11)
Nauseau and/or Vomiting (Gastrointestinal disorders) | 19 (19) | 11 (11)
Dizziness (Nervous system disorders) | 19 (19) | 14 (14)
Rapid Heart Rate (Cardiac disorders) | 18 (18) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/01/NCT03511001/Prot_000.pdf